CLINICAL TRIAL: NCT06918626
Title: INtraoperative Approach With Eventual Clearance of Common bilE Duct by SpyGlass Discover vs Sequential Strategy in Patients With Acute Calculus Cholecystitis and Intermediate/High Risk of Common BiLE Duct Stone
Acronym: INACCESSIBLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Luca Ansaloni, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: INACCESSIBLE
Record Dates: First submitted 2025-03-22; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Acute Calculous Cholecystitiis (ACC)
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients who receive ELC + Spyglass cholangiography (Experimental)
  Interventions: Procedure: ELC + Spyglass cholangiography
- Patients who receive ERCP + Early Laparoscopic cholecystectomy (ELC) in two stage procedures (Active Comparator)
  Interventions: Procedure: ERCP + Early Laparoscopic cholecystectomy (ELC) in two stage procedures

INTERVENTIONS:
Procedure: ELC + Spyglass cholangiography — Study group (Spyglass Discover). Patients will undergo ELC surgery as soon as the ACC diagnosis has been confirmed. During surgery, intra-operative cholangiograpy (IOC) will be performed in order to exclude the presence of CBDS and in case of confirmation or still suspicion of CBDS, the exploration of the common bile duct and its eventual clearance via Spyglass Discover is carried out during ELC.
  Arms: Patients who receive ELC + Spyglass cholangiography
Procedure: ERCP + Early Laparoscopic cholecystectomy (ELC) in two stage procedures — Control group (ELC sequential treatment after possible clearance of CBDS via ERCP). Following the diagnosis of ACC, patients with CBDS high/intermediate risk are introduced either directly, in case of high risk, or after performing second-level diagnostics (MNR cholangiography or endoscopic ultrasound), in the case of intermediate risk, to the ERCP with the aim of eliminating CBDS preoperatively and then the ELC will be performed.
  Arms: Patients who receive ERCP + Early Laparoscopic cholecystectomy (ELC) in two stage procedures

SUMMARY:
INACCESSIBLE trial is a randomized controlled study that compares two different strategies for the treatment of Acute Calculous Cholecystitiis (ACC) patients with high/intermediate risk of CBDS, according to the score by Khoury T (named Israelian Score, IS). If a patient meets the inclusion and exclusion criteria, (s)he will be randomized to receive ERCP + Early Laparoscopic cholecystectomy (ELC) in two stage procedures (control group) or ELC + Spyglass cholangiography (study group). The follow-up will be performed after 30 days and 6 months from intervention with an outpatient medical examination

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of ACC as defined by 2018 Tokyo Guidelines criteria
* have an Israelian Score (IS) for the risk of main bile duct stones of 2 or 3
* be >18 years old
* onset of symptoms ≤7 days before Emergency Department (ED) admission
* provide signed and dated informed consent form
* be willing to comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

* Pregnancy
* Patients unwilling to undergo follow-up assessments
* Patients diagnosed with concomitant cholangitis or pancreatitis
* Acute cholecystitis not related to a gallstone etiology
* Onset of symptoms >7 days before ED admission
* Altered anatomy of the upper gastrointestinal tract due to surgery of the esophagus, stomach and duodenum
* Biliary peritonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-02-18 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Timing of ELC after diagnosis of ACC | At the end of the procedures.
  The rate of patients who perform ELC within 72 hours after ACC diagnosis.

SECONDARY OUTCOMES:
30-day postoperative complication rate according to Clavien Dindo | Day 30
30-day postoperative biliary complication rate | Day 30
30-day postoperative mortality rate | Day 30
Intraoperative complication rate | Day 0
Failure rate of performing the procedure | Day 0
Operative times | Day 0
Conversion to open surgery rate | Day 0
Need of ERCP after in LC + Spyglass cholangiography group | immediately after the procedures, Day 30, 6 months
Postoperative length of stay (PO-LOS) | immediately after the procedures
Total length of stay (T-LOS) | immediately after the procedures
Total readmission rate within 6 months | 6 Months after procedure
Readmission rate within 6 months due to Gallstones Relates Events (GRE) | 6 Months after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia, Italy